CLINICAL TRIAL: NCT06598163
Title: Efficacy of a Digital Health App Five Lives MED to Improve Cognitive Function in Patients With Mild Cognitive Impairment: a Randomised Controlled Trial
Brief Title: Five Lives MED to Improve Cognitive Function in Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SharpTx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FLMED-01
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; cognitive training; computerized cognitive training
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Five Lives MED (Experimental): Participants will use the Five Lives MED app, where they will be offered ~30 min daily sessions including a healthy-habit-forming component and cognitive training.
  They will be able to complete maximum one session per day and will be advised to complete a minimum of 3 sessions per week. The participants can complete more sessions if they wish.
  After each session they have ad-libitum access to the cognitive-training games and educational articles.
  Interventions: Device: Five Lives MED
- Control (No Intervention): Participants in the control group will receive an informational leaflet with up-to-date standard advice on sleep hygiene, diet, and physical exercise, with an explanation on how these relate to brain health.

INTERVENTIONS:
Device: Five Lives MED — Five Lives MED is a mobile application that can be installed on smartphones and tablets using the Android and/or iOS operating systems for use at home.
  The app offers structured sessions that can be completed once per day. Once the session is completed, the app also offers optional access to additional cognitive training exercises and educational articles.
  The intervention sessions begins with a Habit Quest, a physical activity habit building tool delivered through a chat bot. Following the Habit Quest, the participant is guided through a series of gamified cognitive training exercises aimed at improving attention, memory, language and executive function.
  Arms: Five Lives MED

SUMMARY:
The goal of this randomized controlled trial is to determine whether the digital health app Five Lives MED can improve cognitive function in people with mild cognitive impairment (MCI). The main question it aims to answer is:

Can 12 weeks of using Five Lives MED improve global cognitive function in people diagnosed with MCI?

Researchers will compare with a control group who receives a leaflet with standard health information.

Participants in the intervention group will be asked to use the Five Lives MED app 3 times per week at home for 12 weeks.

All participants, in both groups, will undergo cognitive testing and will complete questionnaires at baseline and exit.

DETAILED DESCRIPTION:
Mild cognitive impairment is a significant public health concern. Non-pharmacological interventions, specifically multi-domain lifestyle and computerised cognitive training interventions, offer an accessible, scalable, engaging and potentially effective solution to improve cognitive function.

Five Lives MED is an interventional digital health app consisting of a physical activity habit forming coaching programme and cognitive training exercises.

The purpose of this study is to evaluate the efficacy of the Five Lives MED device; the primary hypothesis is that there is a significant difference in MoCA scores between the intervention group and the control group after the 12-week Five Lives MED intervention, with an effect size of d = 0.50 or greater favouring the intervention group.

This is a multi-centre, randomised, single-blind, controlled study in participants aged ≥ 50 years with mild cognitive impairment. Participants will be randomly assigned to the intervention (Five Lives MED) or control group for a 12-week period on a 1:1 allocation ratio.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mild Cognitive Impairment (also known as mild cognitive disorder [ICD-10-CM; G31.84] or mild neurocognitive disorder (DSM-5)
* Age ≥ 50
* Participant or informant is willing and able to give informed consent for participation in the study
* Ability to read and understand English (UK) or French (France)
* Access to a mobile phone (Apple iOS 12.4 or above or Android 6.0 (Marshmallow) or above) or iPad (Apple iOS 12.4 or above only) with internet connection (mobile or WiFi).

Exclusion Criteria:

* Diagnosis of dementia or evidence of functional impairment inconsistent with MCI
* Severe visual impairment
* Currently undergoing any other cognitive remediation programme
* Currently taking part in any other investigational study that in the opinion of the investigator may impact the data integrity of the current study
* Physical impairment that makes using a mobile device impossible
* Lack of access to an informant
* Participant under guardianship
* Unwilling or unable to tolerate or engage with study procedures
* Physical impairment that makes standing/walking unassisted impossible.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Baseline and Study Exit (12 weeks)
  The pen and paper, full version of the Montreal Cognitive Assessment (MoCA) is a widely used screening tool designed to detect mild cognitive impairment (MCI) and early signs of dementia. It evaluates several cognitive domains, including short-term memory, visuospatial abilities, executive functions, attention, concentration, working memory, language, and orientation to time and place. The MoCA is scored out of 30 points, with a score of 26 or above considered normal. Lower scores indicate potential cognitive impairment, with specific ranges often used to gauge the severity: 18-25 for mild cognitive impairment, 10-17 for moderate cognitive impairment, and below 10 for severe cognitive impairment.

SECONDARY OUTCOMES:
Mild Behavioural Impairment Checklist (MBI-C) | Baseline and Study Exit (12 weeks)
  The Mild Behavioral Impairment Checklist (MBI-C) is a 34-item tool designed to detect the onset of neuropsychiatric symptoms that are significant and persistent, particularly in individuals who are at risk for developing dementia. The MBI-C assesses symptoms across five core domains: decreased motivation, affective dysregulation, impulse control, social inappropriateness, and abnormal perception or thought content. Each item in the checklist is rated based on whether the symptom has been present for at least six months, with severity ratings ranging from mild to severe.
Amsterdam IADL Questionnaire (A-IADL-Q-SV) | Baseline and Study Exit (12 weeks)
  The Amsterdam Instrumental Activities of Daily Living Questionnaire - Short Version (A-IADL-Q-SV) is a concise, informant-based tool designed to assess impairments in instrumental activities of daily living (IADL) in individuals with cognitive decline, including those with dementia. The short version consists of 30 items, covering various daily activities such as household tasks, managing finances, using technology, and leisure activities.
  The total score, or T-score, is normally distributed with a mean of 50 and a standard deviation of 10. The T-score range is approximately 20-80, with higher scores indicating better daily functioning
D-KEFS Trail Making Test | Baseline and Study Exit (12 weeks)
  The Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test is a neuropsychological assessment used to evaluate various aspects of executive functioning, particularly cognitive flexibility, processing speed, and attention. It consists of five conditions that assess visual scanning, number sequencing, letter sequencing, number-letter switching, and motor speed. Each condition has raw and scaled scores, with higher scaled scores indicating better performance.
30-second Chair Stand test (30CST) | Baseline and Study Exit (12 weeks)
  The 30-Second Chair Stand Test (30CST) is a functional fitness test designed to assess lower body strength and endurance, particularly in older adults. The test involves counting how many times an individual can fully stand up from a seated position and sit back down in a chair without using their arms, all within a 30-second period. A higher score indicates better performance. This test is commonly used to evaluate the risk of falls and overall functional mobility in seniors.
Five Lives cognitive tests | Baseline and Study Exit (12 weeks)
  Five Lives offers five digital cognitive tests via iPad or smartphone, each targeting different cognitive functions.
  * the Snap test assesses verbal fluency,
  * the Breeze test measures short-term memory and numerical abilities through word recall tasks,
  * the Cast test evaluates spatial and numerical memory with increasingly complex grid tasks,
  * the Swift test, based on the Stroop Task, measures inhibition by requiring participants to identify the meaning or color of words, and
  * the Twist test assesses processing speed and cognitive control using a digitized version of the Trail Making Test.
  Higher scores indicate better performance.
QoL in Alzheimer's disease (QOL-AD) | Baseline and Study Exit (12 weeks)
  The Quality of Life in Alzheimer's Disease (QOL-AD) scale is a 13-item questionnaire designed to assess the quality of life of individuals diagnosed with Alzheimer's disease from both the patients and informants perspectives. It measures areas such as physical health, mood, relationships, and the ability to perform daily activities. Each item is rated on a 4-point scale from 1 (poor) to 4 (excellent), with total scores ranging from 13 to 52, where higher scores indicate a better perceived quality of life.
Alzheimer's Disease Knowledge Scale (ADKS) | Baseline and Study Exit (12 weeks)
  The Alzheimer's Disease Knowledge Scale (ADKS) is a 30-item true/false questionnaire designed to assess knowledge about Alzheimers disease across several domains, including risk factors, symptoms, diagnosis, treatment, caregiving, and disease progression. Higher scores indicate better knowledge.
International Physical Activity Questionnaire (IPAQ) | Baseline and Study Exit (12 weeks)
  The International Physical Activity Questionnaire (IPAQ) is a widely used self-report tool designed to measure physical activity levels. The IPAQ has been adapted for use with older adults, including those aged 65 and above. The IPAQ can be particularly useful in assessing physical activity levels in this demographic, helping to understand the frequency, intensity, and duration of various types of physical activity, such as walking, moderate, and vigorous activities. Scores will be expressed in metabolic equivalent (MET)-min per week, which higher MET-min indicating more physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Koychev, MD, PhD, Principal Investigator — University of Oxford
Locations (7):
- Hôpital Broca, Service de gériatrie Hôpitaux Universitaire Paris Centre, Université Paris Cité, Paris, Île-de-France Region, France
- United Kingdom (6):
  - Devon Partnership NHS Trust, Exeter, Devon
  - Lancashire & South Cumbria NHS Foundation Trust, Preston, Lancashire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Somerset NHS Foundation Trust, Taunton, Somerset
  - East London NHS Foundation Trust, London
  - South London & Maudsley NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided
The anonymised IPD may be shared with other organisations and researchers, only if the participant has provided informed consent to do so and only if the data is used for other research that has passed ethical approval. Thus, the plan for IPD sharing is currently undecided as it remains to be determined if study audit will be conducted and if future studies will make use of the IPD.

REFERENCES:
- [Background] Gauthier S, Reisberg B, Zaudig M, Petersen RC, Ritchie K, Broich K, Belleville S, Brodaty H, Bennett D, Chertkow H, Cummings JL, de Leon M, Feldman H, Ganguli M, Hampel H, Scheltens P, Tierney MC, Whitehouse P, Winblad B; International Psychogeriatric Association Expert Conference on mild cognitive impairment. Mild cognitive impairment. Lancet. 2006 Apr 15;367(9518):1262-70. doi: 10.1016/S0140-6736(06)68542-5. PMID 16631882
- [Background] Petersen RC. Mild Cognitive Impairment. Continuum (Minneap Minn). 2016 Apr;22(2 Dementia):404-18. doi: 10.1212/CON.0000000000000313. PMID 27042901
- [Background] Jongsiriyanyong S, Limpawattana P. Mild Cognitive Impairment in Clinical Practice: A Review Article. Am J Alzheimers Dis Other Demen. 2018 Dec;33(8):500-507. doi: 10.1177/1533317518791401. Epub 2018 Aug 1. PMID 30068225
- [Background] Sachdev PS, Lipnicki DM, Kochan NA, Crawford JD, Thalamuthu A, Andrews G, Brayne C, Matthews FE, Stephan BC, Lipton RB, Katz MJ, Ritchie K, Carriere I, Ancelin ML, Lam LC, Wong CH, Fung AW, Guaita A, Vaccaro R, Davin A, Ganguli M, Dodge H, Hughes T, Anstey KJ, Cherbuin N, Butterworth P, Ng TP, Gao Q, Reppermund S, Brodaty H, Schupf N, Manly J, Stern Y, Lobo A, Lopez-Anton R, Santabarbara J; Cohort Studies of Memory in an International Consortium (COSMIC). The Prevalence of Mild Cognitive Impairment in Diverse Geographical and Ethnocultural Regions: The COSMIC Collaboration. PLoS One. 2015 Nov 5;10(11):e0142388. doi: 10.1371/journal.pone.0142388. eCollection 2015. PMID 26539987
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Welstead M, Luciano M, Muniz-Terrera G, Taylor AM, Russ TC. Prevalence of Mild Cognitive Impairment in the Lothian Birth Cohort 1936. Alzheimer Dis Assoc Disord. 2021 Jul-Sep 01;35(3):230-236. doi: 10.1097/WAD.0000000000000433. PMID 33480611
- [Background] Gabelle A, Guery M, Doutriaux A, Bettayeb K. Forecasting the Prevalence of Alzheimer's Disease at Mild Cognitive Impairment and Mild Dementia Stages in France in 2022. J Prev Alzheimers Dis. 2023;10(2):259-266. doi: 10.14283/jpad.2023.22. PMID 36946453
- [Background] Vlachos GS, Kosmidis MH, Yannakoulia M, Dardiotis E, Hadjigeorgiou G, Sakka P, Ntanasi E, Stefanis L, Scarmeas N. Prevalence of Mild Cognitive Impairment in the Elderly Population in Greece: Results From the HELIAD Study. Alzheimer Dis Assoc Disord. 2020 Apr-Jun;34(2):156-162. doi: 10.1097/WAD.0000000000000361. PMID 31913961
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol. 1999 Mar;56(3):303-8. doi: 10.1001/archneur.56.3.303. PMID 10190820
- [Background] Tierney MC, Szalai JP, Snow WG, Fisher RH, Nores A, Nadon G, Dunn E, St George-Hyslop PH. Prediction of probable Alzheimer's disease in memory-impaired patients: A prospective longitudinal study. Neurology. 1996 Mar;46(3):661-5. doi: 10.1212/wnl.46.3.661. PMID 8618663
- [Background] Lampit A, Hallock H, Valenzuela M. Computerized cognitive training in cognitively healthy older adults: a systematic review and meta-analysis of effect modifiers. PLoS Med. 2014 Nov 18;11(11):e1001756. doi: 10.1371/journal.pmed.1001756. eCollection 2014 Nov. PMID 25405755
- [Background] Nguyen L, Murphy K, Andrews G. A Game a Day Keeps Cognitive Decline Away? A Systematic Review and Meta-Analysis of Commercially-Available Brain Training Programs in Healthy and Cognitively Impaired Older Adults. Neuropsychol Rev. 2022 Sep;32(3):601-630. doi: 10.1007/s11065-021-09515-2. Epub 2021 Jul 12. PMID 34251578
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Hafdi M, Hoevenaar-Blom MP, Richard E. Multi-domain interventions for the prevention of dementia and cognitive decline. Cochrane Database Syst Rev. 2021 Nov 8;11(11):CD013572. doi: 10.1002/14651858.CD013572.pub2. PMID 34748207
- [Background] Kivipelto M, Mangialasche F, Ngandu T. Lifestyle interventions to prevent cognitive impairment, dementia and Alzheimer disease. Nat Rev Neurol. 2018 Nov;14(11):653-666. doi: 10.1038/s41582-018-0070-3. PMID 30291317
- [Background] Zokaei N, MacKellar C, Cepukaityte G, Patai EZ, Nobre AC. Cognitive Training in the Elderly: Bottlenecks and New Avenues. J Cogn Neurosci. 2017 Sep;29(9):1473-1482. doi: 10.1162/jocn_a_01080. Epub 2016 Nov 29. PMID 27897677
- [Background] Pedulla L, Brichetto G, Tacchino A, Vassallo C, Zaratin P, Battaglia MA, Bonzano L, Bove M. Adaptive vs. non-adaptive cognitive training by means of a personalized App: a randomized trial in people with multiple sclerosis. J Neuroeng Rehabil. 2016 Oct 4;13(1):88. doi: 10.1186/s12984-016-0193-y. PMID 27716336
- [Background] Bodner KA, Goldberg TE, Devanand DP, Doraiswamy PM. Advancing Computerized Cognitive Training for MCI and Alzheimer's Disease in a Pandemic and Post-pandemic World. Front Psychiatry. 2020 Nov 25;11:557571. doi: 10.3389/fpsyt.2020.557571. eCollection 2020. No abstract available. PMID 33329097
- [Background] Costanzo MC, Arcidiacono C, Rodolico A, Panebianco M, Aguglia E, Signorelli MS. Diagnostic and interventional implications of telemedicine in Alzheimer's disease and mild cognitive impairment: A literature review. Int J Geriatr Psychiatry. 2020 Jan;35(1):12-28. doi: 10.1002/gps.5219. Epub 2019 Nov 15. PMID 31617247
- [Background] Zuschnegg J, Schoberer D, Haussl A, Herzog SA, Russegger S, Ploder K, Fellner M, Hofmarcher-Holzhacker MM, Roller-Wirnsberger R, Paletta L, Koini M, Schussler S. Effectiveness of computer-based interventions for community-dwelling people with cognitive decline: a systematic review with meta-analyses. BMC Geriatr. 2023 Apr 12;23(1):229. doi: 10.1186/s12877-023-03941-y. PMID 37041494
- [Background] Chae HJ, Lee SH. Effectiveness of online-based cognitive intervention in community-dwelling older adults with cognitive dysfunction: A systematic review and meta-analysis. Int J Geriatr Psychiatry. 2023 Jan;38(1):e5853. doi: 10.1002/gps.5853. PMID 36468299
- [Background] Li R, Geng J, Yang R, Ge Y, Hesketh T. Effectiveness of Computerized Cognitive Training in Delaying Cognitive Function Decline in People With Mild Cognitive Impairment: Systematic Review and Meta-analysis. J Med Internet Res. 2022 Oct 27;24(10):e38624. doi: 10.2196/38624. PMID 36301590
- [Background] Fiatarone Singh MA, Gates N, Saigal N, Wilson GC, Meiklejohn J, Brodaty H, Wen W, Singh N, Baune BT, Suo C, Baker MK, Foroughi N, Wang Y, Sachdev PS, Valenzuela M. The Study of Mental and Resistance Training (SMART) study-resistance training and/or cognitive training in mild cognitive impairment: a randomized, double-blind, double-sham controlled trial. J Am Med Dir Assoc. 2014 Dec;15(12):873-80. doi: 10.1016/j.jamda.2014.09.010. Epub 2014 Oct 23. PMID 25444575
- [Background] Hagovska M, Olekszyova Z. Impact of the combination of cognitive and balance training on gait, fear and risk of falling and quality of life in seniors with mild cognitive impairment. Geriatr Gerontol Int. 2016 Sep;16(9):1043-50. doi: 10.1111/ggi.12593. Epub 2015 Sep 3. PMID 26338465
- [Background] Ferizaj D, Mavrogenis AF, Tsolaki M, Charisis SK, Drosos GI, Karamitrou I, et al. Effectiveness of mobile computerized cognitive training in adults with mild cognitive impairment: interim analysis of a randomized controlled trial [Preprint]. 2024 Jan 1 [cited 2024 Aug 21]; Available from: https://doi.org/10.21203/rs.3.rs-3099721/v1.
- [Background] Kuster OC, Fissler P, Laptinskaya D, Thurm F, Scharpf A, Woll A, Kolassa S, Kramer AF, Elbert T, von Arnim CA, Kolassa IT. Cognitive change is more positively associated with an active lifestyle than with training interventions in older adults at risk of dementia: a controlled interventional clinical trial. BMC Psychiatry. 2016 Sep 8;16(1):315. doi: 10.1186/s12888-016-1018-z. PMID 27608620
- [Background] Bahar-Fuchs A, Webb S, Bartsch L, Clare L, Rebok G, Cherbuin N, Anstey KJ. Tailored and Adaptive Computerized Cognitive Training in Older Adults at Risk for Dementia: A Randomized Controlled Trial. J Alzheimers Dis. 2017;60(3):889-911. doi: 10.3233/JAD-170404. PMID 28922158
- [Background] Hyer L, Scott C, Atkinson MM, Mullen CM, Lee A, Johnson A, Mckenzie LC. Cognitive Training Program to Improve Working Memory in Older Adults with MCI. Clin Gerontol. 2016 Oct-Dec;39(5):410-427. doi: 10.1080/07317115.2015.1120257. Epub 2016 Mar 2. PMID 29471774
- [Background] Stern Y, Arenaza-Urquijo EM, Bartres-Faz D, Belleville S, Cantilon M, Chetelat G, Ewers M, Franzmeier N, Kempermann G, Kremen WS, Okonkwo O, Scarmeas N, Soldan A, Udeh-Momoh C, Valenzuela M, Vemuri P, Vuoksimaa E; the Reserve, Resilience and Protective Factors PIA Empirical Definitions and Conceptual Frameworks Workgroup. Whitepaper: Defining and investigating cognitive reserve, brain reserve, and brain maintenance. Alzheimers Dement. 2020 Sep;16(9):1305-1311. doi: 10.1016/j.jalz.2018.07.219. Epub 2020 Jan 6. PMID 30222945
- [Background] Chapman SB, Aslan S, Spence JS, Hart JJ Jr, Bartz EK, Didehbani N, Keebler MW, Gardner CM, Strain JF, DeFina LF, Lu H. Neural mechanisms of brain plasticity with complex cognitive training in healthy seniors. Cereb Cortex. 2015 Feb;25(2):396-405. doi: 10.1093/cercor/bht234. Epub 2013 Aug 28. PMID 23985135
- [Background] Kim S, Park E, Cha H, Jung JC, Jung TD, Chang Y. Effects of Cognitive Training in Mild Cognitive Impairmentmeasured by Resting State Functional Imaging. Behav Sci (Basel). 2020 Nov 17;10(11):175. doi: 10.3390/bs10110175. PMID 33213021
- [Background] Demurtas J, Schoene D, Torbahn G, Marengoni A, Grande G, Zou L, Petrovic M, Maggi S, Cesari M, Lamb S, Soysal P, Kemmler W, Sieber C, Mueller C, Shenkin SD, Schwingshackl L, Smith L PhD, Veronese N; European Society of Geriatric Medicine Special Interest Group in Systematic Reviews and Meta-Analyses, Frailty, Sarcopenia, and Dementia. Physical Activity and Exercise in Mild Cognitive Impairment and Dementia: An Umbrella Review of Intervention and Observational Studies. J Am Med Dir Assoc. 2020 Oct;21(10):1415-1422.e6. doi: 10.1016/j.jamda.2020.08.031. PMID 32981668
- [Background] Hu M, Hu H, Shao Z, Gao Y, Zeng X, Shu X, Huang J, Shen S, Wu IXY, Xiao LD, Feng H. Effectiveness and acceptability of non-pharmacological interventions in people with mild cognitive impairment: Overview of systematic reviews and network meta-analysis. J Affect Disord. 2022 Aug 15;311:383-390. doi: 10.1016/j.jad.2022.05.043. Epub 2022 May 18. PMID 35597472
- [Background] Lauenroth A, Ioannidis AE, Teichmann B. Influence of combined physical and cognitive training on cognition: a systematic review. BMC Geriatr. 2016 Jul 18;16:141. doi: 10.1186/s12877-016-0315-1. PMID 27431673
- [Background] Li KZ, Roudaia E, Lussier M, Bherer L, Leroux A, McKinley PA. Benefits of cognitive dual-task training on balance performance in healthy older adults. J Gerontol A Biol Sci Med Sci. 2010 Dec;65(12):1344-52. doi: 10.1093/gerona/glq151. Epub 2010 Sep 13. PMID 20837662
- [Background] Marusic U, Verghese J, Mahoney JR. Cognitive-Based Interventions to Improve Mobility: A Systematic Review and Meta-analysis. J Am Med Dir Assoc. 2018 Jun;19(6):484-491.e3. doi: 10.1016/j.jamda.2018.02.002. Epub 2018 Apr 19. PMID 29680203
- [Background] Karssemeijer EGA, Aaronson JA, Bossers WJ, Smits T, Olde Rikkert MGM, Kessels RPC. Positive effects of combined cognitive and physical exercise training on cognitive function in older adults with mild cognitive impairment or dementia: A meta-analysis. Ageing Res Rev. 2017 Nov;40:75-83. doi: 10.1016/j.arr.2017.09.003. Epub 2017 Sep 12. PMID 28912076
- [Background] Ali N, Tian H, Thabane L, Ma J, Wu H, Zhong Q, Gao Y, Sun C, Zhu Y, Wang T. The Effects of Dual-Task Training on Cognitive and Physical Functions in Older Adults with Cognitive Impairment; A Systematic Review and Meta-Analysis. J Prev Alzheimers Dis. 2022;9(2):359-370. doi: 10.14283/jpad.2022.16. PMID 35543010
- [Background] Gavelin HM, Dong C, Minkov R, Bahar-Fuchs A, Ellis KA, Lautenschlager NT, Mellow ML, Wade AT, Smith AE, Finke C, Krohn S, Lampit A. Combined physical and cognitive training for older adults with and without cognitive impairment: A systematic review and network meta-analysis of randomized controlled trials. Ageing Res Rev. 2021 Mar;66:101232. doi: 10.1016/j.arr.2020.101232. Epub 2020 Nov 26. PMID 33249177
- [Background] Bherer L, Gagnon C, Langeard A, Lussier M, Desjardins-Crepeau L, Berryman N, Bosquet L, Vu TTM, Fraser S, Li KZH, Kramer AF. Synergistic Effects of Cognitive Training and Physical Exercise on Dual-Task Performance in Older Adults. J Gerontol B Psychol Sci Soc Sci. 2021 Sep 13;76(8):1533-1541. doi: 10.1093/geronb/gbaa124. PMID 32803232
- [Background] Montero-Odasso M, Almeida QJ, Burhan AM, Camicioli R, Doyon J, Fraser S, Li K, Liu-Ambrose T, Middleton L, Muir-Hunter S, McIlroy W, Morais JA, Pieruccini-Faria F, Shoemaker K, Speechley M, Vasudev A, Zou GY, Berryman N, Lussier M, Vanderhaeghe L, Bherer L. SYNERGIC TRIAL (SYNchronizing Exercises, Remedies in Gait and Cognition) a multi-Centre randomized controlled double blind trial to improve gait and cognition in mild cognitive impairment. BMC Geriatr. 2018 Apr 16;18(1):93. doi: 10.1186/s12877-018-0782-7. PMID 29661156
- [Background] Bruderer-Hofstetter M, Rausch-Osthoff AK, Meichtry A, Munzer T, Niedermann K. Effective multicomponent interventions in comparison to active control and no interventions on physical capacity, cognitive function and instrumental activities of daily living in elderly people with and without mild impaired cognition - A systematic review and network meta-analysis. Ageing Res Rev. 2018 Aug;45:1-14. doi: 10.1016/j.arr.2018.04.002. Epub 2018 Apr 18. PMID 29679658
- [Background] Joubert C, Chainay H. Aging brain: the effect of combined cognitive and physical training on cognition as compared to cognitive and physical training alone - a systematic review. Clin Interv Aging. 2018 Jul 20;13:1267-1301. doi: 10.2147/CIA.S165399. eCollection 2018. PMID 30057444
- [Background] Zhu X, Yin S, Lang M, He R, Li J. The more the better? A meta-analysis on effects of combined cognitive and physical intervention on cognition in healthy older adults. Ageing Res Rev. 2016 Nov;31:67-79. doi: 10.1016/j.arr.2016.07.003. Epub 2016 Jul 14. PMID 27423932
- [Background] Walton CC, Mowszowski L, Lewis SJ, Naismith SL. Stuck in the mud: time for change in the implementation of cognitive training research in ageing? Front Aging Neurosci. 2014 Mar 17;6:43. doi: 10.3389/fnagi.2014.00043. eCollection 2014. No abstract available. PMID 24672478
- [Background] Gates NJ, Vernooij RW, Di Nisio M, Karim S, March E, Martinez G, Rutjes AW. Computerised cognitive training for preventing dementia in people with mild cognitive impairment. Cochrane Database Syst Rev. 2019 Mar 13;3(3):CD012279. doi: 10.1002/14651858.CD012279.pub2. PMID 30864747
- [Background] Chuang IC, Chiau HY, Liao WW, Wu YR, Chang CH, Wu CY. Effects of computer-based cognitive training combined with physical training for older adults with cognitive impairment: A four-arm randomized controlled trial. Digit Health. 2023 Sep 20;9:20552076231203633. doi: 10.1177/20552076231203633. eCollection 2023 Jan-Dec. PMID 37744745
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Kang M, Ragan BG, Park JH. Issues in outcomes research: an overview of randomization techniques for clinical trials. J Athl Train. 2008 Apr-Jun;43(2):215-21. doi: 10.4085/1062-6050-43.2.215. PMID 18345348
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Carpenter BD, Balsis S, Otilingam PG, Hanson PK, Gatz M. The Alzheimer's Disease Knowledge Scale: development and psychometric properties. Gerontologist. 2009 Apr;49(2):236-47. doi: 10.1093/geront/gnp023. Epub 2009 Mar 25. PMID 19363018
- [Background] Tsang S, Royse CF, Terkawi AS. Guidelines for developing, translating, and validating a questionnaire in perioperative and pain medicine. Saudi J Anaesth. 2017 May;11(Suppl 1):S80-S89. doi: 10.4103/sja.SJA_203_17. PMID 28616007
- [Background] Jutten RJ, Peeters CFW, Leijdesdorff SMJ, Visser PJ, Maier AB, Terwee CB, Scheltens P, Sikkes SAM. Detecting functional decline from normal aging to dementia: Development and validation of a short version of the Amsterdam IADL Questionnaire. Alzheimers Dement (Amst). 2017 Mar 31;8:26-35. doi: 10.1016/j.dadm.2017.03.002. eCollection 2017. PMID 28462387
- [Background] Ismail Z, Aguera-Ortiz L, Brodaty H, Cieslak A, Cummings J, Fischer CE, Gauthier S, Geda YE, Herrmann N, Kanji J, Lanctot KL, Miller DS, Mortby ME, Onyike CU, Rosenberg PB, Smith EE, Smith GS, Sultzer DL, Lyketsos C; NPS Professional Interest Area of the International Society of to Advance Alzheimer's Research and Treatment (NPS-PIA of ISTAART). The Mild Behavioral Impairment Checklist (MBI-C): A Rating Scale for Neuropsychiatric Symptoms in Pre-Dementia Populations. J Alzheimers Dis. 2017;56(3):929-938. doi: 10.3233/JAD-160979. PMID 28059789
- [Background] Chan ATC, Ip RTF, Tran JYS, Chan JYC, Tsoi KKF. Computerized cognitive training for memory functions in mild cognitive impairment or dementia: a systematic review and meta-analysis. NPJ Digit Med. 2024 Jan 3;7(1):1. doi: 10.1038/s41746-023-00987-5. PMID 38172429
- [Background] Irazoki E, Contreras-Somoza LM, Toribio-Guzman JM, Jenaro-Rio C, van der Roest H, Franco-Martin MA. Technologies for Cognitive Training and Cognitive Rehabilitation for People With Mild Cognitive Impairment and Dementia. A Systematic Review. Front Psychol. 2020 Apr 9;11:648. doi: 10.3389/fpsyg.2020.00648. eCollection 2020. PMID 32373018
- [Background] Alnajjar F, Khalid S, Vogan AA, Shimoda S, Nouchi R, Kawashima R. Emerging Cognitive Intervention Technologies to Meet the Needs of an Aging Population: A Systematic Review. Front Aging Neurosci. 2019 Oct 24;11:291. doi: 10.3389/fnagi.2019.00291. eCollection 2019. PMID 31798439
- See also: World Health Organization. Global Status Report on the Public Health Response to Dementia. World Health Organization; 2021. 137 p. — https://www.who.int/publications/i/item/9789240033245